CLINICAL TRIAL: NCT00863252
Title: A Prospective, Randomized, Open Label, Case-Controlled Study on the Efficacy of Mycophenolate Mofetil for IgA Nephropathy Patients With Heavy Proteinuria Despite Angiotensin Blockade
Brief Title: Mycophenolate Mofetil for IgA Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: United Christian Hospital (Other); Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Dr Sydney C.W. Tang, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Roche-ST-01
Record Dates: First submitted 2009-03-15; First posted 2009-03-17 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: IGA Nephropathy
Keywords: proteinuria; creatinine; kidney survival; ESRD
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria; Kidney Failure, Chronic | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MMF
  Interventions: Drug: mycophenolate mofetil
- 2 (Active Comparator): Control
  Interventions: Drug: angiotensin blockade

INTERVENTIONS:
Drug: mycophenolate mofetil — Orally at 0.75 g bd to 1 g bd for 6 months
  Arms: 1
Drug: angiotensin blockade — Continuation of angiotensin blockade
  Arms: 2

SUMMARY:
IgA nephropathy (IgAN) is the commonest primary glomerulonephritis worldwide. In Hong Kong, IgAN accounts for approximately 30% of all primary glomerular diseases, and a significant proportion of young patients (< 50 years of age) on dialysis therapy are sufferers of primary IgAN. To date, no specific therapeutic agent has been consistently shown to halt the progression of IgAN to end-stage renal failure, particularly in patients with persistent significant proteinuria and the presence of chronic tubulointerstitial inflammation on kidney biopsy. In recent years, angiotensin-converting enzyme inhibitors (ACEI) have been found capable of significantly reducing proteinuria in some IgAN patients, while others, particularly those with the ACE DD genotype, showed either absent or unsatisfactory response to angiotensin blockade. Mycophenolate mofetil (MMF) is a marketed immunosuppressive drug which acts by releasing mycophenolic acid (MPA) to inhibit the de novo pathway of purine synthesis, and hence is relatively selective for lymphocytes. Apart from being efficacious for the prophylaxis of renal allograft rejection and for the induction of remission in severe lupus nephritis, MMF has been anecdotally reported to avert progression to allograft failure in recurrent IgAN of the transplanted kidney. Data on the clinical efficacy of MMF in the treatment of primary IgAN, however, is lacking. In the current proposal, we aim to study the clinical efficacy of MMF in patients with biopsy-proven IgAN and clinically significant proteinuria despite angiotensin blockade. Patients will be followed up for at least 5 years to track any survival difference between groups.

DETAILED DESCRIPTION:
(i) STUDY DESIGN

This will be a prospective, randomized, open-label, case-controlled study. Patients of either gender with biopsy-proven IgAN and clinically significant proteinuria despite being on ACEI treatment will be potential candidates (see selection criteria). Eligible patients will be randomized into either of the following groups:

Group I (Intervention arm):

Patients will be given MMF at a daily dose of 1.5 g orally in 2 divided doses in addition to concurrent medications, including ACEI. Duration of therapy is expected to be six months.

Group II (Control arm):

Patient will continue to receive all concurrent medications, including ACEI or angiotensin receptor blocker, at the discretion of the attending renal physician.

(ii) PATIENT SELECTION CRITERIA Inclusion criteria

* Males or females between the ages of 18 and 70 years
* Renal biopsy showing a histological diagnosis IgAN, with predominant or codominant mesangial deposition of IgA on immunofluorescent studies
* Daily urinary protein excretion > 1 g on at least 3 separate occasions
* Serum creatinine < 400 umol/L
* Patients who are willing to give written informed consent and to participate in and comply with the study protocol

Exclusion criteria

* Presence of concomitant glomerular diseases
* Patients with known hypersensitivity to MMF
* Patients receiving treatment with other cytotoxic agents
* Serum creatinine > 400 umol/L
* Women who are lactating, pregnant or of childbearing potential not using, or who are unwilling to use, a reliable contraceptive method during and for 6 weeks following conclusion of MMF therapy. A pregnancy test to exclude pregnancy will be performed for women of childbearing potential prior to recruitment
* Patients who are unable or unwilling to give written informed consent and to participate in and comply with the study protocol
* Presence of systemic infection or malignancy requiring therapy at the time of entry to the study
* Patients simultaneously participating in another study or who have participated in another study within the last 30 days of entry into this study

(iii) PATIENT MONITORING

Patient record

The record of every recruited patient will contain the following information:

* Demographic data
* Medical history including concomitant illness
* All concomitant medications
* Other significant information

Timing of Assessments

All study assessments will be calculated from the date of study entry. The study follow-up schedule will be as follows:

* Baseline, then
* Two-weekly for the first month, then
* Monthly for the 2nd - 6th month, at the end of which MMF will be withdrawn, then
* Three-monthly until at least 5 years of follow up

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 70 years
* Renal biopsy showing a histological diagnosis IgAN, with predominant or codominant mesangial deposition of IgA on immunofluorescent studies
* Daily urinary protein excretion > 1 g on at least 3 separate occasions
* Serum creatinine < 400 umol/L
* Patients who are willing to give written informed consent and to participate in and comply with the study protocol

Exclusion Criteria:

* Presence of concomitant glomerular diseases
* Patients with known hypersensitivity to MMF
* Patients receiving treatment with other cytotoxic agents
* Serum creatinine > 400 umol/L
* Women who are lactating, pregnant or of childbearing potential not using, or who are unwilling to use, a reliable contraceptive method during and for 6 weeks following conclusion of MMF therapy. A pregnancy test to exclude pregnancy will be performed for women of childbearing potential prior to recruitment
* Patients who are unable or unwilling to give written informed consent and to participate in and comply with the study protocol
* Presence of systemic infection or malignancy requiring therapy at the time of entry to the study
* Patients simultaneously participating in another study or who have participated in another study within the last 30 days of entry into this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-03; Primary Completion 2004-06 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
24 hour urinary protein excretion | 18 months to 5 years

SECONDARY OUTCOMES:
Renal survival Serum creatinine level and creatinine clearance Urine albumin-to-creatinine ratio | at least 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sydney CW Tang, MD, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine and Geriatrics, United Christian Hospital, Hong Kong, China

REFERENCES:
- [Result] Tang S, Leung JC, Chan LY, Lui YH, Tang CS, Kan CH, Ho YW, Lai KN. Mycophenolate mofetil alleviates persistent proteinuria in IgA nephropathy. Kidney Int. 2005 Aug;68(2):802-12. doi: 10.1111/j.1523-1755.2005.00460.x. PMID 16014059